CLINICAL TRIAL: NCT02479802
Title: Pilot Study on the Effects of Plasma Exchange on Motor Dysfunction and Cognitive Function in Patients With Amyotrophic Lateral Sclerosis
Brief Title: Efficacy and Safety of Plasma Exchange With Albumin in Patients With Amyotrophic Lateral Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Biologicals, LLC (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IG1309
Record Dates: First submitted 2015-06-10; First posted 2015-06-24 (Estimated); Results first posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: plasma exchange; albumin
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Albumin (Experimental): Plasma exchange with Albumin
  Interventions: Biological: Albumin

INTERVENTIONS:
Biological: Albumin — 27 plasma exchange procedures using Albumin 5% (estimated 3000 mL per plasma exchange) as replacement solution:
  * three weeks of intensive treatment with two plasma exchanges per week
  * twenty-one weeks of maintenance treatment with one weekly plasma exchange
  Other Names: Human Albumin 5%; Albutein 5%

SUMMARY:
Pilot, phase II, prospective, open-label, uncontrolled study of plasma exchange with 5% albumin in 10 subjects having a definite, possible, or probable diagnosis of Amyotrophic Lateral Sclerosis (ALS).

ELIGIBILITY:
Inclusion Criteria:

* Signed written-informed consent.
* Subjects over 18 years of age, and less than 70 years old.
* Subjects with a definite, possible, or probable diagnosis of ALS, according to the revised El Escorial criteria.
* Subjects having experienced their first ALS symptoms within 18 months before recruitment/consent.
* FVC > 70%
* Subjects must be medically suitable for study participation and of complying with all planned aspects of the protocol including blood sampling at the time of inclusion in the study.

Exclusion Criteria:

* Subjects with a clinically significant preexisting lung disease not attributable to ALS.
* Subjects with a diagnosis of other neurodegenerative diseases or diseases associated with dysfunction of the motor neurons that can confuse the diagnosis of ALS.
* Participation in other clinical trials, or the reception of any other investigational drug in the six months prior to the start of the study.
* Female subjects who are pregnant, currently breastfeeding, or attempting to conceive during the study.
* Difficult peripheral venous access precluding plasma exchange and inability to implement a viable alternative catheter to make continued performing plasma exchange visits according to protocol
* Any contraindication for plasma exchange or abnormal coagulation parameters according clinical criteria from apheresis team
* A history of frequent adverse reactions (serious or otherwise) to blood products.
* Hypersensitivity to albumin or allergies to any of the components of Albutein.
* Subjects that can not interrupt treatment with acetylsalicylic acid or oral anticoagulants
* Plasma creatinine > 2mg/dl.
* Present a history of heart disease including ischemic heart disease or congestive heart failure.
* Presence of prior conduct disorders requiring pharmacologic intervention, with less than 3 months of stable treatment
* Any condition that complicates adherence to study protocol (illness with less than one year of expected survival, drug or alcohol abuse, etc.)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

REFERENCES:
- [Derived] Povedano M, Paipa A, Barcelo M, Woodward MK, Ortega S, Dominguez R, Aragones ME, Horrillo R, Costa M, Paez A. Plasma exchange with albumin replacement and disease progression in amyotrophic lateral sclerosis: a pilot study. Neurol Sci. 2022 May;43(5):3211-3221. doi: 10.1007/s10072-021-05723-z. Epub 2021 Nov 18. PMID 34791571

RESULTS

PARTICIPANT FLOW:
Groups:
- Albumin: Plasma exchange with Albumin
  Albumin: 27 plasma exchange procedures using Albumin 5% (estimated 3000 mL per plasma exchange) as replacement solution:
  * three weeks of intensive treatment with two plasma exchanges per week
  * twenty-one weeks of maintenance treatment with one weekly plasma exchange
Period: Overall Study
Arm/Group | Albumin
Started | 13
Completed | 11
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Albumin
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (9.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Spain | 13

OUTCOME MEASURES:

1. Primary Outcome: Changes From Baseline in the Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R)
Description: Amyotrophic Lateral Sclerosis Functional Rating Scale-Revised (ALSFRS-R) includes 12 questions classified into 3 subdomains: bulbar function (3 questions), fine and gross motor skills (6 questions), and respiratory function (3 questions) to assess the level self sufficiency. Each task was graded according to a 5-point scale from 0 (incapable) to 4 (normal ability) with a total score from 0 (worst) to 48 (best).
Time Frame: Baseline, Weeks 4, 12, 25, 36, and 48
Population: Two subjects discontinued from the study early.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Albumin
Number analyzed (Participants) | 13
units on a scale
  Week 4 | -1.0 [-1.0 to 0.0]
  Week 12: number analyzed (Participants) | 12
  Week 12 | -1.5 [-4.0 to 0.0]
  Week 25: number analyzed (Participants) | 11
  Week 25 | -4.0 [-8.0 to -3.0]
  Week 36: number analyzed (Participants) | 10
  Week 36 | -5.5 [-9.0 to -3.0]
  Week 48: number analyzed (Participants) | 11
  Week 48 | -10.0 [-14.0 to -7.0]
Statistical Analysis 1: Comparison: Albumin; Change from Baseline at Week 48; Test type: Other; p < 0.0001, t-test, 1 sided

2. Primary Outcome: Changes From Baseline in Percent Predicted Forced Vital Capacity (FVC)
Time Frame: Baseline, Weeks 4, 12, 25, 36, and 48
Population: Two subjects discontinued from the study.
Measure: Median (Inter-Quartile Range); unit: percentage of predicted value
Arm/Group | Albumin
Number analyzed (Participants) | 13
percentage of predicted value
  Week 4 | -6.0 [-9.0 to 2.0]
  Week 12: number analyzed (Participants) | 12
  Week 12 | -3.5 [-12.5 to 0.0]
  Week 25: number analyzed (Participants) | 11
  Week 25 | -9.0 [-23.0 to -6.0]
  Week 36: number analyzed (Participants) | 9
  Week 36 | -12.0 [-22.0 to -12.0]
  Week 48: number analyzed (Participants) | 11
  Week 48 | -23.0 [-38.0 to -9.0]
Statistical Analysis 1: Comparison: Albumin; Change from Baseline at Week 48; Test type: Other; p = 0.0006, t-test, 1 sided

3. Secondary Outcome: Changes From Baseline in ALS Cognitive Function Determined by the ALS-Cognitive Behavioral Screen (ALS-CBS) Test
Description: ALS-CBS test is composed of 2 sections. The first section of the ALS-CBS test includes a questionnaire completed by the caregiver regarding behavior and symptoms status. It is comprised of 15 questions inquiring about possible changes over time in participant's behavior that the caregiver has noticed since the onset of ALS symptoms. Each item is scored on a scale ranging from 0 (worst) to 3 (best) yielding a total 0= large changes to 45=no changes. There were 4 additional questions related to current behavioral symptoms (depression, anxiety, fatigue, and emotional liability). Each question was scored as 0= the presence of symptoms and 1= no current symptoms, giving a total score between 0 and 4. The second section of the ALB-CBS test is for cognitive screening and consists of four items: attention, concentration, follow-up and monitoring, and initiation and recovery. These items were scored 0-5 with a maximum score of 20 (0= cognitive impairment, 20= no apparent cognitive impairment).
Time Frame: Baseline, Weeks 25 and 48
Population: Two subjects discontinued from the study.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Albumin
Number analyzed (Participants) | 11
units on a scale
  Behavior Status Week 25 | 0.0 [-3.0 to 2.0]
  Behavior Status Week 48 | -1.0 [-6.0 to 1.0]
  Symptom Status Week 25 | 0.0 [-1.0 to 1.0]
  Symptom Status Week 48 | 0.0 [-1.0 to 1.0]
  Cognitive Screening Week 25 | 0.0 [-2.0 to 1.0]
  Cognitive Screening Week 48 | -1.0 [-3.0 to 2.0]

4. Secondary Outcome: Motor Evoked Potential in Thenar and Hypothenar Eminence, and Anterior Tibialis Muscle
Description: Surface electromyography was performed to record motor evoked potential in the distal muscles of the upper limbs (thenar and hypothenar eminence) and dorsiflexor muscles of the lower limbs (anterior tibialis) after electrical stimulation.
Time Frame: Baseline, Weeks 4, 12, 25, 36, and 48
Population: Two subjects were discontinued from the study.
Measure: Median (Inter-Quartile Range); unit: mV
Arm/Group | Albumin
Number analyzed (Participants) | 13
mV
  Right Tibialis Anterior Week 0: number analyzed (Participants) | 12
  Right Tibialis Anterior Week 0 | 2.6 [0.5 to 6.2]
  Right Tibialis Anterior Week 4 | 4.9 [1.5 to 7.1]
  Right Tibialis Anterior Week 12: number analyzed (Participants) | 12
  Right Tibialis Anterior Week 12 | 3.1 [0.6 to 5.5]
  Right Tibialis Anterior Week 25: number analyzed (Participants) | 11
  Right Tibialis Anterior Week 25 | 1.9 [0.4 to 4.5]
  Right Tibialis Anterior Week 36: number analyzed (Participants) | 10
  Right Tibialis Anterior Week 36 | 2.1 [0.3 to 5.5]
  Right Tibialis Anterior Week 48: number analyzed (Participants) | 11
  Right Tibialis Anterior Week 48 | 1.2 [0.0 to 3.2]
  Left Tibialis Anterior Week 0: number analyzed (Participants) | 12
  Left Tibialis Anterior Week 0 | 3.2 [1.2 to 6.6]
  Left Tibialis Anterior Week 4 | 3.1 [0.4 to 5.3]
  Left Tibialis Anterior Week 12: number analyzed (Participants) | 12
  Left Tibialis Anterior Week 12 | 3.3 [0.1 to 5.2]
  Left Tibialis Anterior Week 25: number analyzed (Participants) | 11
  Left Tibialis Anterior Week 25 | 2.6 [0.1 to 4.3]
  Left Tibialis Anterior Week 36: number analyzed (Participants) | 10
  Left Tibialis Anterior Week 36 | 2.1 [0.2 to 4.1]
  Left Tibialis Anterior Week 48: number analyzed (Participants) | 11
  Left Tibialis Anterior Week 48 | 1.0 [0.0 to 3.7]
  Right Thenar Eminence (APB) Week 0: number analyzed (Participants) | 12
  Right Thenar Eminence (APB) Week 0 | 4.0 [0.6 to 9.4]
  Right Thenar Eminence (APB) Week 4 | 4.4 [0.6 to 7.3]
  Right Thenar Eminence (APB) Week 12: number analyzed (Participants) | 12
  Right Thenar Eminence (APB) Week 12 | 3.0 [0.9 to 4.1]
  Right Thenar Eminence (APB) Week 25: number analyzed (Participants) | 11
  Right Thenar Eminence (APB) Week 25 | 2.6 [0.4 to 3.7]
  Right Thenar Eminence (APB) Week 36: number analyzed (Participants) | 9
  Right Thenar Eminence (APB) Week 36 | 1.2 [0.4 to 3.4]
  Right Thenar Eminence (APB) Week 48: number analyzed (Participants) | 11
  Right Thenar Eminence (APB) Week 48 | 0.6 [0.1 to 3.1]
  Left Thenar Eminence (APB) Week 0 | 6.4 [1.4 to 8.7]
  Left Thenar Eminence (APB) Week 4: number analyzed (Participants) | 12
  Left Thenar Eminence (APB) Week 4 | 2.6 [0.9 to 6.2]
  Left Thenar Eminence (APB) Week 12: number analyzed (Participants) | 11
  Left Thenar Eminence (APB) Week 12 | 3.1 [0.6 to 6.4]
  Left Thenar Eminence (APB) Week 25: number analyzed (Participants) | 10
  Left Thenar Eminence (APB) Week 25 | 1.9 [0.2 to 6.0]
  Left Thenar Eminence (APB) Week 36: number analyzed (Participants) | 10
  Left Thenar Eminence (APB) Week 36 | 0.6 [0.2 to 2.7]
  Left Thenar Eminence (APB) Week 48: number analyzed (Participants) | 11
  Left Thenar Eminence (APB) Week 48 | 0.5 [0.2 to 1.2]
  Right Hypothenar Eminence (ADM) Week 0: number analyzed (Participants) | 11
  Right Hypothenar Eminence (ADM) Week 0 | 6.4 [0.6 to 8.1]
  Right Hypothenar Eminence (ADM) Week 4 | 7.4 [6.3 to 7.9]
  Right Hypothenar Eminence (ADM) Week 12: number analyzed (Participants) | 12
  Right Hypothenar Eminence (ADM) Week 12 | 5.8 [2.7 to 8.1]
  Right Hypothenar Eminence (ADM) Week 25: number analyzed (Participants) | 10
  Right Hypothenar Eminence (ADM) Week 25 | 5.1 [2.6 to 5.8]
  Right Hypothenar Eminence (ADM) Week 36: number analyzed (Participants) | 10
  Right Hypothenar Eminence (ADM) Week 36 | 5.0 [2.8 to 6.1]
  Right Hypothenar Eminence (ADM) Week 48: number analyzed (Participants) | 11
  Right Hypothenar Eminence (ADM) Week 48 | 3.2 [0.6 to 6.9]
  Left Hypothenar Eminence (ADM) Week 0: number analyzed (Participants) | 12
  Left Hypothenar Eminence (ADM) Week 0 | 6.2 [3.3 to 8.8]
  Left Hypothenar Eminence (ADM) Week 4: number analyzed (Participants) | 12
  Left Hypothenar Eminence (ADM) Week 4 | 5.5 [3.5 to 8.2]
  Left Hypothenar Eminence (ADM) Week 12: number analyzed (Participants) | 11
  Left Hypothenar Eminence (ADM) Week 12 | 4.4 [2.1 to 7.4]
  Left Hypothenar Eminence (ADM) Week 25: number analyzed (Participants) | 11
  Left Hypothenar Eminence (ADM) Week 25 | 3.8 [1.1 to 6.5]
  Left Hypothenar Eminence (ADM) Week 36: number analyzed (Participants) | 10
  Left Hypothenar Eminence (ADM) Week 36 | 4.0 [0.2 to 7.0]
  Left Hypothenar Eminence (ADM) Week 48: number analyzed (Participants) | 11
  Left Hypothenar Eminence (ADM) Week 48 | 2.4 [0.4 to 7.3]

5. Secondary Outcome: Changes From Baseline in Amyotrophic Lateral Sclerosis Assessment Questionnaire 40 (ALSA-Q40).
Description: The Amyotrophic Lateral Sclerosis Assessment Questionnaire 40 (ALSA-40) consists of 40 items grouped into 5 representative dimensions associated with quality of life. The first 4 scales (physical mobility, activities of daily living, food and drink, communication) refer to deficits and subsequent disabilities as a result of the disease. The fifth scale (emotional functioning) reflects how the subject is facing his/her physical deterioration emotionally. Each item is scored from 0 to 4 according to a gradation of symptom onset frequency (never, rarely, sometimes, often, and always). From raw scores, an index from 0 to 100 is obtained for each dimension, which allow comparisons to be made with the other dimensions as well as a straightforward interpretation of results (0 = better state of health as measured by the questionnaire; 100 = poorer state of health).
Time Frame: Baseline, Weeks 25 and 48
Population: Two subject discontinued from the study early.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Albumin
Number analyzed (Participants) | 11
units on a scale
  Physical Mobility Week 25 | 10.0 [0.0 to 20.0]
  Physical Mobility Week 48 | 32.5 [7.5 to 50.0]
  ADL/Independence Week 25 | 12.5 [-2.5 to 45.0]
  ADL/Independence Week 48 | 25.0 [7.5 to 45.0]
  Eating and Drinking Week 25 | 0.0 [0.0 to 25.0]
  Eating and Drinking Week 48 | 8.3 [0.0 to 58.3]
  Communication Week 25 | 0.0 [0.0 to 28.6]
  Communication Week 48 | 0.0 [0.0 to 35.7]
  Emotional Functioning Week 25 | 5.0 [-2.5 to 22.5]
  Emotional Functioning Week 48 | 7.5 [0.0 to 20.0]

6. Secondary Outcome: Percentage of Plasma Exchange Sessions Associated With One Adverse Event or Adverse Reaction, Including Clinically Significant Changes in Vital Signs or Lab Parameters
Time Frame: During the Treatment Phase (24 weeks)
Measure: Mean (Standard Deviation); unit: percentage of PE sessions
Units Other Than Participants: Number of PE sessions
Arm/Group | Albumin
Number analyzed (Participants) | 13
Number analyzed (Number of PE sessions) | 330
percentage of PE sessions | 0.9 (2.22)

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study (48 weeks).
Arm/Group | Albumin
All-Cause Mortality (participants affected / at risk) | 1/13
Serious Adverse Events (participants affected / at risk) | 4/13
Other Adverse Events (participants affected / at risk) | 12/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albumin (N=13)
Pneumonia (Infections and infestations) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Albumin (N=13)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 6 (6)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Chest injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Weight decreased (Investigations) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 3 (3)
Presyncope (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Mechanical ventilation (Surgical and medical procedures) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No